CLINICAL TRIAL: NCT03561909
Title: An Open-label, Single Centre, Exploratory Trial Investigating the Kinetics of Platelets Transfused to Healthy, Male Subjects
Brief Title: Kinetics of Blood Platelets Transfused to Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prophylix Pharma AS (Industry)
Collaborators: Larix A/S (Industry); Fraunhofer Institute for Translational Medicine and Pharmacology ITMP (Other); Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other); Bioscientia Central Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PX-0
Record Dates: First submitted 2018-06-04; First posted 2018-06-19 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Fetal and Neonatal Alloimmune Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune | interventions — Platelet Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet transfusion (Other): HLA-A2 and/or HLA A9 negative healthy study subjects will be transfused with a small dose of platelets from an HLA-A2 and/or HLA-A9 positive donor.
  Interventions: Other: Platelet transfusion

INTERVENTIONS:
Other: Platelet transfusion — Transfusion of a platelet dose from 20 × 10ˆ9 to 100 × 10ˆ9.

SUMMARY:
The current phase 0 trial is preceding the phase 1/2 trial of a newly developed drug, NAITgam, for the prevention of fetal and neonatal alloimmune thrombocytopenia (FNAIT) - a rare, but potentially very severe bleeding condition in the fetus or newborn. FNAIT may occur in women whose blood platelets do not express HPA-1a. If the fetus has inherited HPA-1a from the father, the mother's immune system may be stimulated to produce HPA-1a antibodies if HPA-1a positive fetal blood platelets enter the maternal circulation during delivery. In a subsequent pregnancy, such antibodies will cross the placenta and may reduce the number of HPA-1a positive blood platelets in the fetus, which in turn may result in severe bleeding in the fetus or newborn.

The phase 1/2 study of NAITgam will examine NAITgam's ability to eliminate HPA-1a positive blood platelets that has been transfused to healthy male subjects, whose blood platelet do not express HPA-1a. The ability to quickly eliminate transfused HPA-1a positive platelets is considered as a surrogate endpoint for NAITgam's ability to prevent formation of antibodies against HPA-1a after delivery of an HPA-1a positive child.

The current phase 0 trial will examine the survival of blood platelets transfused to healthy male individuals without subsequent administration of NAITgam. The natural survival of transfused platelet, as determined in the phase 0 trial, will be compared with the survival of transfused HPA-1a positive platelets after administration of NAITgam in the phase 1/2 trial. The aim of the phase 0 trial is first, to determine the dose of blood platelet that should be transfused to the healthy subjects in the phase 1/2 trial; and secondly, to determine the optimal time point, after transfusion of platelets, for administration of NAITgam in the phase 1/2 trial.

Eight to 24 healthy male subjects will be included in the phase 0 trial. After transfusion of platelets, blood samples will be collected at regular intervals to determine the proportion of transfused blood platelets. Differences between tissue type antigens between donor and recipient will be used to determine the proportion of transfused platelets. Survival of transfused platelets will be performed by flow cytometry - a method that can be used to quantify very small proportions of cells in the blood. Fluorochrome-conjugated monoclonal antibodies against HLA-A2 and HLA-A9 will be used for flow cytometric identification the transfused platelets.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any trial related procedures are performed
2. Healthy, male subjects
3. Age ≥18 and < 50 years old
4. BMI < 30kg/mˆ2
5. HLA-A2 and/or HLA-A9 negative

Exclusion Criteria:

1. History of hypersensitivity to platelet concentrates or human plasma protein
2. Subjects with known IgA deficiency and anti-IgA antibodies
3. Blood donation received within 3 weeks
4. Platelet counts < 150 × 10ˆ9/L or > 450 × 10ˆ9/L
5. Any type of known platelet function disorder
6. Treatment with non-steroidal anti-inflammatory drugs (NSAIDs, e.g. acetylsalicylic acid) or selective serotonin reuptake inhibitors within 7 days prior to Visit 1
7. Chronic or ongoing active infectious disease requiring systemic treatment including, but not limited to, chronic and renal infection, chronic chest infection with bronchiectasis, and tuberculosis
8. Participation in any other interventional clinical trial during the trial period
9. Subjects known or suspected of not being able to comply with this trial protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
10. Presence of HLA-antibodies class I (MFI level > 3000)
11. Signs of previous or ongoing infection with HIV and/or Hepatitis B and/or C virus

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Terminal elimination half live | The terminal elimination half live of transfused platelets will be determined based on the survival of platelets within the first 5 days after trandfusion
  Determination of the terminal elimination half live of a single platelet dose transfused to healthy male subjects

SECONDARY OUTCOMES:
Cmax | Will be determined within the first 5 days after transfusion
  The peak platelet concentration
AUC | Will be determined within the first 5 days after transfusion
  The area under the platelet concentration versus time curve
Clearance | Will be determined within the first 5 days after transfusion
  Natural clearance of platelets from the circulation

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kjeldsen-Kragh, MD, PhD, Study Chair — Prophylix Pharma AS; Michaela Köhm, MD, Principal Investigator — Fraunhofer Institute for Molecular Biology and Applied Ecology IME
Locations (1):
- Fraunhofer Institute for Molecular Biology and Applied Ecology IME, Frankfurt am Main, Hessia, Germany

IPD SHARING:
Plan to Share IPD: No